CLINICAL TRIAL: NCT04740190
Title: Combination Talazoparib - Carboplatin for Recurrent High-grade Glioma With DNA Damage Repair Deficiency (DDRd)
Brief Title: Talazoparib - Carboplatin for Recurrent High-grade Glioma With DDRd
Acronym: TAC-GReD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW-20396
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Glioma; Recurrent Glioblastoma; Poly ADP Ribose Polymerase (PARP) Inhibitor; PTEN Gene Inactivation; IDH Mutation
Keywords: recurrent glioblastoma; recurrent glioma; PARP inhibitor; IDH mutation; PTEN gene inactivation; BRCAness; DNA Damage Repair Deficiency
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — talazoparib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- interventional arm (Experimental): Single fraction, low dose (2Gy) whole brain radiation therapy, followed by combination talazoparib and carboplatin
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — low dose whole brain radiation, followed by combination talazoparib and carboplatin
  Other Names: Carboplatin; whole brain irradiation

SUMMARY:
In view of the strong biological rationale of employing PARP inhibition in high grade glioma, the current study purposes testing of talazoparib in a biomarker-enriched group of glioma. Carboplatin will be added to sensitize the tumor to PARP inhibition, and low dose radiation therapy will be applied to increase talazoparib drug penetration through blood-brain barrier. The goal is to estimate the effect size of such combinational treatment approach in recurrent high-grade glioma with DNA damage repair deficiency (dDDR)

DETAILED DESCRIPTION:
Recurrent high grade glioma with dDDR, defined by genomic aberrations associated including IDH mutation, PTEN mutation and "BRCAness" signature as defined by next-generation-sequencing (NGS) based comprehensive genomic profiling, will be enrolled.

Patients will receive treatment in 7-day cycle. D1-4: Oral talazoparib 0.75mg daily; D1: Carboplatin (AUC 1.5). On cycle 1 day 1 low dose whole radiation radiation therapy will be given to increase drug penetration. Primary outcome is 6-month progression free survival (PFS-6) by RANO criteria. The study intended to recruit 33 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven diagnosis of WHO grade 3-4 glioma
2. Tumor with one or more putatively pathogenic mutations or homozygous deletion in the genes associated with DDR or genomic instability, as listed below, will be eligible for the study. Genetic analysis on tumor tissue should be performed with next-generation-sequencing (NGS) based analysis to screen for the following genomic aberrations, which included,

   1. IDH mutation
   2. PTEN mutation
   3. "BRCAness" signature (ATM, ATR, BAP1, BRCA1, BRCA2, CDK12, CHEK1, CHEK2, FANCA, FANCC, FANCD2, FANCE, FANCF, PALB2, NGS1, WRN, RAD50, RAD51B, RAD51C, RAD51D, MRE11A, BLM, BRIP1) The molecular profiling results will be considered eligible for screening only if they are performed in laboratories accredited by the College of American Pathologists (CAP) and certified to meet Clinical Laboratory Improvement Amendments (CLIA).
3. Patients will be eligible if the original histology was lower-grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma is made.
4. Patients who did not have recent surgery for their glioblastoma must have shown unequivocal radiographic evidence for tumor progression by contrast-enhanced MRI scan (or CT scan for patients with non-compatible devices) within 21 days prior to registration. Patients who did have surgery with a post-operative contrast-enhanced scan falling outside the 5-week window prior to registration, must have a repeat MRI scan (or CT scan for patients with non-compatible devices) within 21 days prior to registration.
5. Patients must have passed an interval of 6 months or greater between completion of prior radiotherapy and registration. If patients have not passed an interval of at least 6 months, they may still be eligible if they meet one or more of the following criteria:

   1. New areas of tumor outside the original radiotherapy fields as determined by the investigator, or
   2. Histologic confirmation of tumor through biopsy or resection, or
   3. Nuclear medicine imaging, MR spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than radiation necrosis obtained within 28 days of registration AND an interval of at least 90 days between completion of radiotherapy and registration.
6. Patients unable to undergo MR imaging because of non-compatible devices can be enrolled provided CT scans are obtained and are of sufficient quality. Patients without non-compatible devices may not use CT scans performed to meet this requirement.
7. Prior history of standard dose CNS radiation of 50-60Gy in 25-30 fractions, or 40Gy in 15 Fractions.
8. Patients must have recovered from the toxic effects of prior therapy, and there must be a minimum time of 28 days prior to registration from the administration of any investigational agent or prior cytotoxic therapy with the following exceptions:

   1. 14 days from administration of vincristine
   2. 42 days from administration of nitrosoureas
   3. 21 days from administration of procarbazine
9. Patients having undergone recent resection of their high-grade glioma (within 5 weeks prior to registration) must have recovered from the effects of surgery. For CNS related core or needle biopsies, a minimum of 7 days must have elapsed prior to registration.
10. Residual disease following resection of recurrent glioblastoma is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a post- operative or intra-operative MRI scan (or CT scan for patients with non-compatible devices) must be performed prior to registration.
11. At least 18 years of age.
12. World Health Organisation (WHO) performance status 0-2 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks
13. Normal bone marrow and organ function as defined below:

    1. Marrow: Hemoglobin ≥10.0 gm/dL, absolute granulocyte count (AGC) ≥1,000/mm3 platelets ≥100,000/mm3, absolute lymphocyte count ≥1000/mm3.
    2. Hepatic: Serum/plasma total bilirubin ≤1.5 x upper limit of normal (ULN) with the exception of <2.9 mg/dL for patients with Gilbert's disease, ALT (SGPT) and AST (SGOT) ≤2.5 x ULN.
    3. Renal: Serum/plasma creatinine (sCr) ≤1.5 x upper limit of normal, or creatinine clearance (CrCl) ≥50 mL/min.
    4. Serum/plasma albumin > 3.0 gm/dL
14. For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 5 months after the last dose of study treatments. Such methods include: combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
15. Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

1. Prior therapy with PARP inhibitor
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1 year (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
3. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
   2. Transmural myocardial infarction within the last 6 months prior to registration
   3. History of stroke or transient ischemic attack within 6 months prior to registration.
   4. Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically
   5. Significant peripheral vascular disease.
   6. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   7. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring
   8. Hospitalization or precluding study therapy at the time of registration
   9. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function other than screening panel and
   10. Coagulation parameters are not required for entry into this protocol.
   11. Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Progression free survival in 6 months | 6 month
  Free from disease progression based on RANO criteria

SECONDARY OUTCOMES:
Overall survival | 1 year
  from date of study enrollment to the date of death from any cause
Objective response rate | 1 year
  The percentage of patients with radiologically complete or partial response as determined by the investigator according to RANO criteria
Duration of response | 1 year
  The time interval between the time patient develops radiologically complete or partial response to disease progression according to RANO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Aya Helali, MD, PhD, Principal Investigator — Department of Clinical Oncology
Locations (1):
- Department of Clinical Oncology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No